CLINICAL TRIAL: NCT06366217
Title: Efficacy of the MydCombi on Pupillary Dilation in Pediatric and Adult Patients
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 20-32530A
Record Dates: First submitted 2024-04-10; First posted 2024-04-15 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Dilation; Pupil Reaction Absent
MeSH Terms: conditions — Dilatation, Pathologic; Pupil Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- MydCombi (Experimental): Patients will be dilated using MydCombi drug: (tropicamide 1% and phenylephrine HCl 2.5%) ophthalmic spray in one eye for a few seconds once
  Interventions: Device: MydCombi Device; Drug: MydCombi Drug
- Standard of Care (No Intervention): Participants will receive the standard of care dilation: tropicamide 1% and phenylephrine 2.5%

INTERVENTIONS:
Device: MydCombi Device — ophthalmic spray
  Arms: MydCombi
Drug: MydCombi Drug — Tropicamide 1% and phenylephrine HCl 2.5%
  Arms: MydCombi

SUMMARY:
To raise the standard of care, improve the overall patient experience and streamline practice flow, Eyenovia has developed an innovative mydriatic to be delivered as a microdose by a specialized dispenser. While still achieving effective pupil dilation, MydCombi has the potential to increase patient throughput at practicing offices by decreasing time spent eye dropping patients, eliminating time wasted waiting between drop instillations and ensuring more accurate drug delivery. The proposed study hopes to demonstrate the non-inferiority of using MydCombi to achieve pupillary dilation in patients compared to standard of care eye drops.

DETAILED DESCRIPTION:
The proposed study strives to demonstrate the non-inferiority of using MydCombi to achieve pupillary dilation in patients compared to standard-of-care (SOC) eye drops in a randomized trial.

Primary Aim: Demonstrate non-inferiority of using MydCombi to achieve pupillary dilation compared to standard-of-care eye drops in patients.

Participants 2 years or older undergoing standard pupillary dilation will be randomized to use MydCombi in one eye and standard of care pupillary dilation in another eye.

ELIGIBILITY:
Inclusion Criteria:

* Receiving pupillary dilation in both eyes as part of the participant's standard of care.

Exclusion Criteria:

* Pupillary or anterior segment abnormality
* Participants with pre-existing health conditions that would prevent pupillary dilation.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-09-30 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Percent change in Spherical equivalent | Before dilation and 30 minutes after dilation
  Cycloplegia is the paralysis of the ciliary muscle of the eye resulting in dilatation of the pupil and paralysis of accommodation.
  Cycloplegia is defined as the "change score." Change scores were calculated by subtracting the spherical equivalent value after dilation from the value before dilation for each eye.
Percent Change in maximum pupil diameter | Before dilation and 30 minutes after dilation
  The pupil is the opening in the center of the iris (the structure that gives particpant's eyes their color). The diameter is a straight line passing from side to side through the center of the pupil, which is shaped like a circle.
Percent Change in pupil constriction percentage | Before and 30 minutes after dilation
  Pupillary constriction percentage was calculated by the pupillometer in response to a 180-micro watt flash: (maximum - minimum) / maximum

SECONDARY OUTCOMES:
Percent Change in Intraocular Pressure | Before and 30 minutes After Dilation
  Intraocular pressure is the pressure, or force, inside of the participants eyes. Specifically, it's a measurement of the fluid pressure in the participant's aqueous humor.

CONTACTS AND LOCATIONS:
Overall Officials: Julius Oatts, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No